CLINICAL TRIAL: NCT00072709
Title: A Randomized, Double-Blind, Placebo-Controlled, Stratified, Parallel-Group, Multicenter, Dose-Ranging Study Evaluating Four Oral Doses of TCH346 (1.0, 2.5, 7.5 and 15 mg) Administered Once Daily in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study Evaluating TCH346 and Placebo Administered Once Daily in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTCH346A2211
Record Dates: First submitted 2003-11-07; First posted 2003-11-11 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — dibenzo(b,f)oxepin-10-ylmethyl-methyl-prop-2-ynyl-amine

INTERVENTIONS:
Drug: TCH346

SUMMARY:
This is a global multicenter study designed to evaluate the safety and clinical effects of 4 oral doses of TCH346 (1.0, 2.5, 7.5, and 15 mg) compared to placebo in patients with mild or mild to moderate stages of ALS. The study consists of 3 phases: screening (up to 2 weeks), run-in (16 weeks), and a double-blind treatment phase of variable duration (at least 24 weeks).

ELIGIBILITY:
Inclusion criteria:

* clinical diagnosis of laboratory-supported probable, probable, or definite ALS;
* sporadic or familial ALS;
* ALS symptom onset for no more than 3 yrs at study entry;
* FVC equal to or more than 70%;
* patients who are either riluzole naive or patients who are receiving concomitant treatment with riluzole at a stable dose of riluzole (50 mg bid) at study start.

Exclusion criteria:

* Known or suspected chronic infectious disease including HIV, hepatitis B, or hepatitis C.
* Clinically significant ECG abnormalities.
* Known hypersensitivity to study drug or related drugs (e.g. selegiline, MAO-A and B inhibitors, or tricyclic antidepressants).
* Patients treated with potent inhibitors of CYP1A2 or CYP3A4 (a list of such inhibitors will be provided to the investigator).
* Treatment with MAO-A and B inhibitors (including selegiline) within the past 30 days.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2003-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Rate of functional decline as defined by the ALS Functional Rating Scale-Revised

SECONDARY OUTCOMES:
Survival time
Functional outcome measures including pulmonary function and manual muscle strength assessments (every visit except screening)
Neurocognitive evaluation in a subset of patients(every visit except screening)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis USA, East Hanover, New Jersey, United States
- Novartis Belgium, Vilvoorde, Belgium
- Novartis CANADA, Dorval, Quebec, Canada
- Novartis France, Rueil-Malmaison, France
- Novartis Germany, Nuremberg, Germany
- Novartis Italy, Saronno, Italy
- Novartis Netherlands, Arnhem, Netherlands
- Novartis Switzerland, Bern, Switzerland
- Novartis UK, Frimley, United Kingdom